CLINICAL TRIAL: NCT04250935
Title: The Relationship Between Neurocognitive Changes and Brain-Induced Neurotrophic Factor Levels in Patients Undergoing Coronary Artery Bypass Surgery
Brief Title: Brain-Induced Neurotrophic Factor Levels in Patients Undergoing Coronary Artery Bypass Surgery
Status: Completed | Type: Observational
Sponsor: Bozok University (Other)
Responsible Party: Principal Investigator, Ökkeş Hakan Miniksar, Asist.Prof., Bozok University
Other Study IDs: 20194466
Record Dates: First submitted 2020-01-30; First posted 2020-01-31 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Cognitive Dysfunction
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Patients with cognitive dysfunction — Mini Mental Test Those with a score below 21 points

SUMMARY:
In patients undergoing coronary artery bypass surgery, the relationship between neurocognitive changes seen in the early period and brain-induced neurotrophic factor serum levels will be investigated.

DETAILED DESCRIPTION:
Although postoperative cognitive dysfunction (POKD) is the most common neurological complication in patients undergoing coronary artery bypass grafting (CABG) surgery, its pathophysiology is still not fully understood. However, the quality of this dysfunction has not been properly measured. In addition to clinical tests, biomarkers are often used to detect the presence of POKD. In this study, it was aimed to evaluate the relationship between intraoperative and postoperative brain-derived neurotrophic factor serum levels and POKD in patients undergoing CABG surgery.

This prospective observational study is planned to include 30 adult patients aged 40-90 years. Patients with stroke history, neurodegenerative disease, seizure history, alcohol use, general anxiety, hearing deficit, unilateral carotid artery stenosis greater than 70%, and carotid artery bilateral stenosis greater than 50% will be excluded from the study.

This study aimed to determine perioperative changes in serum brain-derived neurotrophic factor levels in patients undergoing CABG surgery.

ELIGIBILITY:
Inclusion Criteria:

* At Least Primary School Graduates,
* Not Using Drugs That May Affect Cognitive Functions,
* No Alcohol Substance Use,
* Without Psychiatric And Neurological Diseases

Exclusion Criteria:

* Uneducated Patients,
* Drug Users Who May Affect Cognitive Functions (Antipsychotic, Antidepressant),
* Have Alcohol And Substance Use Disorders,
* Those With A History Of Central Nervous System Disease That May Cause Cognitive Dysfunction (Such As Stroke, Neurodegenerative Disease, Seizure, General Anxiety),
* Hearing Deficit,
* Patients With Unilateral Carotid Artery Stenosis Greater Than 70% And Bilateral Stenosis Greater than 50% Carotid Artery

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Volunteer patients to be included in the study: 30 adult patients who will undergo coronary artery bypass grafting (CABG) surgery
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Postoperative cognitive dysfunction | 4 days
  Relationship between serum brain-derived neurotrophic factor level and cognitive dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Yozgat Bozok University Research Hospital, Study Director — Yozgat
Locations (1):
- Bozok University Medical Center, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Can be announced after the work is completed.

REFERENCES:
- [Derived] Miniksar OH, Cicekcioglu F, Kilic M, Honca M, Miniksar DY, Gocmen AY, Kacmaz O, Oz H. Decreased brain-derived neurotrophic factor levels may predict early perioperative neurocognitive disorder in patients undergoing coronary artery bypass surgery: A prospective observational pilot study. J Clin Anesth. 2021 Aug;71:110235. doi: 10.1016/j.jclinane.2021.110235. Epub 2021 Mar 25. PMID 33774438